CLINICAL TRIAL: NCT05661630
Title: THE EFFECT OF SEX EDUCATION AND COUNSELING GIVEN TO WOMEN WITH STOMIA WITH EX-PLISSIT MODEL ON SEXUAL QUALITY OF LIFE AND SEXUAL LIFE SATISFACTION
Brief Title: THE EFFECT OF SEX EDUCATION AND COUNSELING GIVEN TO WOMEN WITH STOMIA WITH THE EX-PLISSIT MODEL ON SEXUAL LIFE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: NESLİHAN YILMAZ SEZER (Other)
Responsible Party: Sponsor-Investigator, NESLİHAN YILMAZ SEZER, Faculty of Nursing, Ankara University
Organization: Ankara University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 18/173
Record Dates: First submitted 2022-12-14; First posted 2022-12-22 (Actual); Last update posted 2022-12-22 (Actual); Status verified 2022-12

CONDITIONS: Stoma Colostomy; Stoma Ileostomy
MeSH Terms: interventions — Educational Status; Counseling

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EX-PLISSIT (Experimental)
  Interventions: Other: EDUCATION AND COUNSELING WITH EX-PLISSIT MODEL
- CONTROL (No Intervention)

INTERVENTIONS:
Other: EDUCATION AND COUNSELING WITH EX-PLISSIT MODEL — In addition to the routine procedure, the women in the experimental group of the research will be given sexual education and counseling with the EX-PLISSIT model. The steps to be followed in accordance with this model are as follows; Session 1 Permission Limited Information The Specific Suggestions The IT-Intensive Therapy Session 2 At the beginning of the interview, the data forms will be reapplied, and then the homework given in the first session will be discussed. The information that the patient needs in line with his questions will be given within the steps of the Ex-PLISSIT model, within the steps of allowing, limited information, special recommendations and, if necessary, intensive therapy.
  Session 3 At the beginning of the interview, the data forms will be applied for the last time and the patient's questions, if any, will be answered and the session will be ended.
  Arms: EX-PLISSIT

SUMMARY:
In this study, it was aimed to determine the effect of sexual education and counseling given to women with stoma with the Ex-PLISSIT model on their sexual life quality and sexual life satisfaction.

H1: Female patients with permanent stoma who were given sexual education and counseling with the EX-PLISSIT model had a higher quality of life score measured by the Sexual Quality of Life scale.

H2: Female patients with permanent stoma who were given sexual education and counseling with the EX-PLISSIT model had higher mean scores of sexual life satisfaction.

ELIGIBILITY:
Inclusion Criteria for Research

* Permanent stoma for at least 6 months
* Not receiving active surgical treatment, chemotherapy and radiotherapy (at least 6 previous treatments have been completed)
* Married
* Agreeing to participate in the research and obtaining written permission,
* Over 18 years Research Exclusion Criteria
* Using antidepressants or using sedatives
* Having a diagnosed psychiatric problem,
* Women with diagnosed sexual dysfunction will not be included in the study. Exclusion Criteria from Research
* Do not complete the study,
* Surgical treatment, radiotherapy or chemotherapy started due to an urgent necessity during the working process, Patients who die during the study will be excluded.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2023-01-02 (Estimated); Primary Completion 2023-12-29 (Estimated); Study Completion 2023-12-29 (Estimated)

PRIMARY OUTCOMES:
Change in Sexual Life Quality | at the beginning of the study, 1 month later and 3 months later
  The scale is easy to apply, 6-point Likert type, which individuals can answer on their own, and consists of 18 items. Each item is expected to be answered considering the sexual life in the last four weeks. Each item of the scale is scored between 1 and 6. The items of the scale are scored as "I totally agree"=1, "I strongly agree"=2, "I partially agree"=3, "I partially disagree"=4, "I strongly disagree"=5, "I strongly disagree"=6 and 1 Questions 5, 9, 13 and 18 are reverse coded. The range of points that can be obtained from the scale is between 18-108.
Change in satisfaction with sexual life | at the beginning of the study, 1 month later and 3 months later
  VAS is a 10-cm-long measurement tool. The left end of the scale reads "I am not satisfied at all" and the right end reads "very satisfied". A high score on the scale indicated a high level of satisfied and a score of 0 pointed to no satisfied.
Change in satisfaction with marital relationship | at the beginning of the study, 1 month later and 3 months later
  VAS is a 10-cm-long measurement tool. The left end of the scale reads "I am not satisfied at all" and the right end reads "very satisfied". A high score on the scale indicated a high level of satisfied and a score of 0 pointed to no satisfied.

IPD SHARING:
Plan to Share IPD: Undecided